CLINICAL TRIAL: NCT00372151
Title: The Value of Augmenting L-Theanine in the Management of Schizophrenia: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: L-Theanine in the Management of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sha'ar Menashe Mental Health Center (Other)
Collaborators: Stanley Medical Research Institute (Other); Beersheva Mental Health Center (Other Government)
Responsible Party: Michael S Ritsner, Technion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Theanine 10/2006.ctil
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizoaffective disorders; Theonine; Augmentation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — theanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-Theanine (Experimental)
  Interventions: Dietary Supplement: L-Theanine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Theanine — 400 mg/day, caps.
  Arms: L-Theanine
Other: Placebo — caps.
  Arms: Placebo

SUMMARY:
The aim of the proposed study is to investigate the efficacy and safety of add-on gamma-glutamylethylamide (L-theanine) versus a placebo for antipsychotic treatment for 8 weeks in a randomized, double-blind, parallel group study of 60 patients with schizophrenia and schizoaffective disorders.

DETAILED DESCRIPTION:
This is a two-year randomized placebo-controlled double-blind investigation of the use of augmentative L-theanine in the management of 60 patients with schizophrenia and schizoaffective disorders. We will investigate several outcome variables in these patients including the positive and negative symptoms, affective features, emotional distress, neuropsychological testing, side effects, and the quality of life. Participating subjects on stable antipsychotic treatment will be randomized to receive for 8 weeks either L-theanine (400 mg/day) or a placebo in addition to regular ongoing antipsychotic medication for 8 weeks. Subjects will be assessed at baseline and after 2, 4, 6, and 8 weeks of treatment using psychiatric rating scales, self-reported questionnaires, and a neuropsychological battery of tests. The efficacy and safety of augmenting antipsychotic treatment with L-theanine will be analyzed.

The Cambridge Neuropsychological Test Automated Battery (CANTAB) will be administered at commencement and completion of the study. The CANTAB battery consists of a series of interrelated computerized tests of visual and movement skills, attention and memory, and executive function, administered via a touch sensitive screen. The nonverbal nature of the CANTAB tests makes them largely language independent and culture free. These tests are run on an IBM-compatible personal computer with a touch-sensitive screen. Neuropsychological testing lasts approximately 2 hours. Subjects complete the tests in a fixed order with a break half-way through the testing session. For a description of the nature of these tests, the performance measures used, and how the test scores are derived, see (http://www.cantab.com/cantab/site/home.acds). The neuropsychological tests are categorized onto five cognitive domains: visual and movement skills, attention, memory, learning, sustained attention, and executive function: Motor Screening, Big/Little Circle, Reaction Time, Matching to Sample Visual Search, Delayed Matching to Sample, Pattern Recognition Memory, Spatial Recognition Memory, Spatial Span, Rapid visual information processing, Spatial working memory, Intra/Extra Dimensional Set Shift, and Stockings of Cambridge. In addition to raw scores from these tasks, the average value of the z-scores of the CANTAB neurocognitive tasks will be used to determine cognitive indices in specific domains.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, men or women
* DSM-IV criteria for schizophrenia or schizoaffective disorder
* At least 4 on the Clinical Global Impression Scale
* At least two weeks of ongoing treatment with current antipsychotic agents.
* Ability and willingness to sign an informed consent form for participation in the study.

Exclusion Criteria:

* Evidence of serious neurologic or endocrine disorder, for example severe head trauma, seizure disorder, dementia, Cushings disease, or thyroid disorder, mental retardation, alcohol or drug abuse.
* Renal disease
* Hepatic dysfunction
* Pregnant women
* Patients receiving mood stabilizing medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The Clinical Global Impression Scale | every two weeks
The Positive and Negative Syndrome Scale | every two weeks
The Scale for the Assessment of Negative Symptoms | every two weeks
The Calgary Depression Scale for Schizophrenia | every two weeks
The Hamilton Scale for Anxiety | every two weeks
Cambridge Neuropsychological Test Automated Battery (CANTAB) | every 4 weeks

SECONDARY OUTCOMES:
The Global Assessment of Functioning | every two weeks
The Talbieh Brief Distress Inventory | every two weeks
The State/Trait Anxiety Inventory | every two weeks
The Quality of Life Scale | every two weeks
The Quality of Life Enjoyment and Satisfaction Questionnaire | every two weeks
The Extrapyramidal Symptom Rating Scale | every two weeks
Barnes Akathisia Scale | every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Ritsner, MD, PhD, Principal Investigator — Sha'ar Menashe Mental Health Center; Yael Ratner, MD, Study Director — Sha'ar Menashe Mental Health Center; Anatoly Gibel, MD, Study Director — Sha'ar Menashe Mental Health Center; Chanoch Miodownik, MD, Study Director — Be'er Sheva Mental Health Center; Tatyana Shleifer, MD, Study Director — Be'er Sheva Mental Health Center
Locations (2):
- Israel (2):
  - Be'er Sheva Mental Health Center, Beersheba
  - Sha'ar Menashe Mental Health Center, Hadera

REFERENCES:
- [Background] Yamada T, Terashima T, Okubo T, Juneja LR, Yokogoshi H. Effects of theanine, r-glutamylethylamide, on neurotransmitter release and its relationship with glutamic acid neurotransmission. Nutr Neurosci. 2005 Aug;8(4):219-26. doi: 10.1080/10284150500170799. PMID 16493792
- [Background] Yokogoshi H, Terashima T. Effect of theanine, r-glutamylethylamide, on brain monoamines, striatal dopamine release and some kinds of behavior in rats. Nutrition. 2000 Sep;16(9):776-7. doi: 10.1016/s0899-9007(00)00384-1. No abstract available. PMID 10978861
- [Derived] Miodownik C, Maayan R, Ratner Y, Lerner V, Pintov L, Mar M, Weizman A, Ritsner MS. Serum levels of brain-derived neurotrophic factor and cortisol to sulfate of dehydroepiandrosterone molar ratio associated with clinical response to L-theanine as augmentation of antipsychotic therapy in schizophrenia and schizoaffective disorder patients. Clin Neuropharmacol. 2011 Jul-Aug;34(4):155-60. doi: 10.1097/WNF.0b013e318220d8c6. PMID 21617527
- [Derived] Ritsner MS, Miodownik C, Ratner Y, Shleifer T, Mar M, Pintov L, Lerner V. L-theanine relieves positive, activation, and anxiety symptoms in patients with schizophrenia and schizoaffective disorder: an 8-week, randomized, double-blind, placebo-controlled, 2-center study. J Clin Psychiatry. 2011 Jan;72(1):34-42. doi: 10.4088/JCP.09m05324gre. Epub 2010 Nov 30. PMID 21208586